CLINICAL TRIAL: NCT02445989
Title: Effects of Contraceptive Ring on Vaginal Microbiota, HIV Shedding and Local Immunity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeanne Marrazzo, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 48663; R01HD077872 (NIH)
Record Dates: First submitted 2015-04-20; First posted 2015-05-15 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Bacterial Vaginosis; HIV
Keywords: HIV; Contraceptive Vaginal Ring; Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclic NuvaRing CVR Use (Active Comparator): CVR use for 3 weeks, remove for 1 week, then replace
  Interventions: Drug: NuvaRing
- Continuous NuvaRing CVR Use (Experimental): CVR use for 4 weeks, then replace
  Interventions: Drug: NuvaRing

INTERVENTIONS:
Drug: NuvaRing — Provide NuvaRing to women seeking contraception
  Other Names: Contraceptive vaginal ring

SUMMARY:
The investigators propose to explore the hypothesis-supported by limited data-that a contraceptive vaginal ring (CVR) that is commonly used in the United States, the NuvaRing, will enhance women's genital and reproductive health. The investigators propose that this CVR will increase the bacteria that help the vaginal environment protect against infection by HIV and other STIs, and that in women who already have HIV, use of the CVR will lower the quantity of HIV that is shed in the female genital tract.

DETAILED DESCRIPTION:
The investigators objective is to study effects of a contraceptive vaginal ring (CVR) containing estrogen and progesterone (NuvaRing) on vaginal bacteria, HIV shedding, and local immunity in women. The investigators will build on data that support a favorable effect of CVR on vaginal bacteria. Bacterial vaginosis (BV) is found in >50% of women in sub-Saharan Africa. BV significantly increases risk of HIV acquisition in, and HIV transmission to male partners from, HIV-infected women, genital HIV shedding, and viral set point in infected male partners. Pregnancy is also an independent risk for HIV acquisition and transmission. Contraception comprises critical biomedical prevention for women with or at risk for HIV. Systemic depot progesterone-commonly used throughout Africa-may independently increase risk of HIV acquisition and transmission. Hormonal interventions preventing unintended pregnancy and promoting a protective vaginal microenvironment could synergistically reduce HIV risk especially combined with topical antiretrovirals (ARV). The investigators propose NuvaRing use may contribute to reduction in BV, pregnancy prevention, and decreased rates of HIV shedding in HIV-infected women. Sustained vaginal delivery of contraceptive and ARV PrEP as "multicomponent prevention" is a major focus for scientists but effects on the vaginal environment need careful definition before broad implementation.

Total duration of follow up is no more than 8 months, with 5 months of CVR usage.

ELIGIBILITY:
Inclusion Criteria:

* BV+ by Amsel Criteria
* Not intending to become pregnant over the course of the study
* If HIV infected, not taking ART
* Capable of providing written informed consent

Exclusion Criteria:

* Current pregnancy
* Desire/intent to become pregnant over the course of the study
* Contraindications to hormonal contraceptive use
* Current cigarette smoking if age is older than 35 years
* Unable to comprehend consent material because of language barrier or psychological difficulty

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Quantity of L. crispatus determined by species-specific qPCR assay | Up to 8 months

SECONDARY OUTCOMES:
Rates of bacterial vaginosis during contraceptive ring uses | Up to 8 months
Number of adverse events with CVR use | Up to 8 months
Acceptability of CVR to male sex partners of study participants assessed by questionnaire | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Marrazzo, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Thika Clinic, Thika, Kenya

REFERENCES:
- [Background] Polis CB, Curtis KM. Use of hormonal contraceptives and HIV acquisition in women: a systematic review of the epidemiological evidence. Lancet Infect Dis. 2013 Sep;13(9):797-808. doi: 10.1016/S1473-3099(13)70155-5. Epub 2013 Jul 19. PMID 23871397
- [Background] van der Straten A, Montgomery ET, Cheng H, Wegner L, Masenga G, von Mollendorf C, Bekker L, Ganesh S, Young K, Romano J, Nel A, Woodsong C. High acceptability of a vaginal ring intended as a microbicide delivery method for HIV prevention in African women. AIDS Behav. 2012 Oct;16(7):1775-86. doi: 10.1007/s10461-012-0215-0. PMID 22644068
- [Background] Kiser PF, Johnson TJ, Clark JT. State of the art in intravaginal ring technology for topical prophylaxis of HIV infection. AIDS Rev. 2012 Jan-Mar;14(1):62-77. PMID 22297505
- [Background] Marrazzo JM, Martin DH, Watts DH, Schulte J, Sobel JD, Hillier SL, Deal C, Fredricks DN. Bacterial vaginosis: identifying research gaps proceedings of a workshop sponsored by DHHS/NIH/NIAID. Sex Transm Dis. 2010 Dec;37(12):732-44. doi: 10.1097/OLQ.0b013e3181fbbc95. PMID 21068695
- [Background] Atashili J, Poole C, Ndumbe PM, Adimora AA, Smith JS. Bacterial vaginosis and HIV acquisition: a meta-analysis of published studies. AIDS. 2008 Jul 31;22(12):1493-501. doi: 10.1097/QAD.0b013e3283021a37. PMID 18614873
- [Background] Cohen CR, Lingappa JR, Baeten JM, Ngayo MO, Spiegel CA, Hong T, Donnell D, Celum C, Kapiga S, Delany S, Bukusi EA. Bacterial vaginosis associated with increased risk of female-to-male HIV-1 transmission: a prospective cohort analysis among African couples. PLoS Med. 2012;9(6):e1001251. doi: 10.1371/journal.pmed.1001251. Epub 2012 Jun 26. PMID 22745608
- [Background] Veres S, Miller L, Burington B. A comparison between the vaginal ring and oral contraceptives. Obstet Gynecol. 2004 Sep;104(3):555-63. doi: 10.1097/01.AOG.0000136082.59644.13. PMID 15339769
- [Background] Ahrendt HJ, Nisand I, Bastianelli C, Gomez MA, Gemzell-Danielsson K, Urdl W, Karskov B, Oeyen L, Bitzer J, Page G, Milsom I. Efficacy, acceptability and tolerability of the combined contraceptive ring, NuvaRing, compared with an oral contraceptive containing 30 microg of ethinyl estradiol and 3 mg of drospirenone. Contraception. 2006 Dec;74(6):451-7. doi: 10.1016/j.contraception.2006.07.004. Epub 2006 Sep 27. PMID 17157101
- [Background] Mugo NR, Heffron R, Donnell D, Wald A, Were EO, Rees H, Celum C, Kiarie JN, Cohen CR, Kayintekore K, Baeten JM; Partners in Prevention HSV/HIV Transmission Study Team. Increased risk of HIV-1 transmission in pregnancy: a prospective study among African HIV-1-serodiscordant couples. AIDS. 2011 Sep 24;25(15):1887-95. doi: 10.1097/QAD.0b013e32834a9338. PMID 21785321
- [Background] Taha TE, James MM, Hoover DR, Sun J, Laeyendecker O, Mullis CE, Kumwenda JJ, Lingappa JR, Auvert B, Morrison CS, Mofensen LM, Taylor A, Fowler MG, Kumenda NI, Eshleman SH. Association of recent HIV infection and in-utero HIV-1 transmission. AIDS. 2011 Jul 17;25(11):1357-64. doi: 10.1097/QAD.0b013e3283489d45. PMID 21572305
- [Background] Heffron R, Donnell D, Rees H, Celum C, Mugo N, Were E, de Bruyn G, Nakku-Joloba E, Ngure K, Kiarie J, Coombs RW, Baeten JM; Partners in Prevention HSV/HIV Transmission Study Team. Use of hormonal contraceptives and risk of HIV-1 transmission: a prospective cohort study. Lancet Infect Dis. 2012 Jan;12(1):19-26. doi: 10.1016/S1473-3099(11)70247-X. Epub 2011 Oct 3. PMID 21975269
- [Background] Mugwanya K, Baeten JM, Mugo NR, Irungu E, Ngure K, Celum C. High-dose valacyclovir HSV-2 suppression results in greater reduction in plasma HIV-1 levels compared with standard dose acyclovir among HIV-1/HSV-2 coinfected persons: a randomized, crossover trial. J Infect Dis. 2011 Dec 15;204(12):1912-7. doi: 10.1093/infdis/jir649. Epub 2011 Oct 12. PMID 21998479
- [Background] Marrazzo JM, Thomas KK, Fiedler TL, Ringwood K, Fredricks DN. Relationship of specific vaginal bacteria and bacterial vaginosis treatment failure in women who have sex with women. Ann Intern Med. 2008 Jul 1;149(1):20-8. doi: 10.7326/0003-4819-149-1-200807010-00006. PMID 18591634
- [Background] Baeten JM, Kahle E, Lingappa JR, Coombs RW, Delany-Moretlwe S, Nakku-Joloba E, Mugo NR, Wald A, Corey L, Donnell D, Campbell MS, Mullins JI, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Genital HIV-1 RNA predicts risk of heterosexual HIV-1 transmission. Sci Transl Med. 2011 Apr 6;3(77):77ra29. doi: 10.1126/scitranslmed.3001888. PMID 21471433